CLINICAL TRIAL: NCT00420212
Title: A Randomized, Multicenter, Double-Blind, Placebo-Controlled, Dose-Comparison Study to Determine the Efficacy and Safety of BG00012 in Subjects With Relapsing-Remitting Multiple Sclerosis
Brief Title: Efficacy and Safety of Oral BG00012 in Relapsing-Remitting Multiple Sclerosis
Acronym: DEFINE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 109MS301
Record Dates: First submitted 2007-01-08; First posted 2007-01-11 (Estimated); Results first posted 2014-06-02 (Estimated); Last update posted 2015-01-26 (Estimated); Status verified 2015-01

CONDITIONS: Relapsing-Remitting Multiple Sclerosis
Keywords: relapsing; oral; remitting; multiple sclerosis
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Recurrence; Multiple Sclerosis | interventions — Dimethyl Fumarate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo (Placebo Comparator): Participants received two placebo capsules orally three times daily (TID)
  Interventions: Drug: Placebo
- BG00012 240 mg Twice Daily (BID) (Experimental): Participants received two 120 mg BG00012 capsules orally twice daily (BID) and two placebo capsules orally once daily (QD)
  Interventions: Drug: BG00012
- BG00012 240 mg 3 Times Daily (TID) (Experimental): Participants received two 120 mg BG00012 capsules orally three times daily (TID)
  Interventions: Drug: BG00012

INTERVENTIONS:
Drug: BG00012
  Other Names: dimethyl fumarate; Tecfidera®
  Arms: BG00012 240 mg 3 Times Daily (TID); BG00012 240 mg Twice Daily (BID)
Drug: Placebo
  Arms: Placebo

SUMMARY:
To determine if treatment with BG00012 can decrease the number of MS relapses during a certain time period. To determine if, over time, BG00012 treatment can decrease the number of certain types of brain lesions commonly seen in MS patients and slow down the time it takes for the disease to get worse.

The purpose of this study is also to determine the safety of BG00012 and how well it is tolerated. Another goal is to see what effect BG00012 may have on tests and evaluations used to assess MS.

ELIGIBILITY:
Key Inclusion Criteria:

* Unless otherwise specified, to be eligible to participate in this study, candidates must meet the following eligibility criteria at the time of the randomization:
* Must have a confirmed diagnosis of RRMS according to McDonald criteria #1-4.
* Must have a baseline EDSS between 0.0 and 5.0, inclusive.
* Must have relapsing-remitting disease course.

Key Exclusion Criteria:

* Unless otherwise specified, candidates will be excluded from study entry if any of the following exclusion criteria exist at randomization:
* Other chronic disease of the immune system, malignancies, acute urologic, pulmonary, gastrointestinal disease.
* Pregnant or nursing women.

Note: Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1234 (Actual)
Dates: Start 2007-01; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (159):
- United States (39):
  - Research Site, Gilbert, Arizona
  - Research Site, Phoenix, Arizona
  - Research Site, San Francisco, California
  - Research Site, New Haven, Connecticut
  - Research Site, Washington D.C., District of Columbia
  - Research Site, Vero Beach, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Evanston, Illinois
  - Research Site, Palos Heights, Illinois
  - Research Site, Fort Wayne, Indiana
  - Research Site, Indianapolis, Indiana
  - Research Site, Des Moines, Iowa
  - Research Site, Wichita, Kansas
  - Research Site, Lexington, Kentucky
  - Research Site, Brighton, Massachusetts
  - Research Site, Hopedale, Massachusetts
  - Research Site, Lexington, Massachusetts
  - Research Site, Springfield, Massachusetts
  - Research Site, Worcester, Massachusetts
  - Research Site, Farmington Hills, Michigan
  - Research Site, Minneapolis, Minnesota
  - Research Site, Columbia, Missouri
  - Research Site, St Louis, Missouri
  - Research Site, Henderson, Nevada
  - Research Site, Las Vegas, Nevada
  - Research Site, Lebanon, New Hampshire
  - Research Site, Albany, New York
  - Research Site, Staten Island, New York
  - Research Site, Raleigh, North Carolina
  - Research Site, Dayton, Ohio
  - Research Site, Erie, Pennsylvania
  - Research Site, Hershey, Pennsylvania
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, East Providence, Rhode Island
  - Research Site, Providence, Rhode Island
  - Research Site, San Antonio, Texas
  - Research Site, Newport News, Virginia
  - Research Site, Wien, Virginia
  - Research Site, Seattle, Washington
- Australia (9):
  - Research Site, Camperdown, New South Wales
  - Research Site, Chatswood, New South Wales
  - Research Site, Fitzroy
  - Research Site, Geelong
  - Research Site, Heidelberg
  - Research Site, Kogarah
  - Research Site, Liverpool
  - Research Site, Melbourne
  - Research Site, Newcastle
- Austria (4):
  - Research Site, Vienna, Vienna
  - Research Site, Graz
  - Research Site, Innsbruck
  - Research Site, Linz
- Belgium (8):
  - Research Site, Antwerp
  - Research Site, Bruges
  - Research Site, Charleroi
  - Research Site, Diepenbeek
  - Research Site, Leuven
  - Research Site, Lommel
  - Research Site, Sijsele-Damme
  - Research Site, Woluwe
- Research Site, Banja Luka, Republic of Srpksa, Bosnia and Herzegovina
- Canada (7):
  - Research Site, Burnaby, British Columbia
  - Research Site, Halifax, Nova Scotia
  - Research Site, Ottawa, Ontario
  - Research Site, Lévis, Quebec
  - Research Site, Québec, Quebec
  - Research Site, Regina, Saskatchewan
  - Research Site, Montreal
- Research Site, Zagreb, Croatia
- Czechia (7):
  - Research Site, Brno
  - Research Site, Jihlava
  - Research Site, Opava
  - Research Site, Ostrava
  - Research Site, Pilsen
  - Research Site, Prague
  - Research Site, Teplice
- France (4):
  - Research Site, Clermont-Ferrand
  - Research Site, Nice
  - Research Site, Paris
  - Research Site, Rennes
- Germany (15):
  - Research Site, Bad Neustadt-Saale
  - Research Site, Berlin
  - Research Site, Bochum
  - Research Site, Düsseldorf
  - Research Site, Essen
  - Research Site, Gieben
  - Research Site, Halle
  - Research Site, Hamburg
  - Research Site, Hanover
  - Research Site, Leipzig
  - Research Site, Minden
  - Research Site, München
  - Research Site, Münster
  - Research Site, Osnabrück
  - Research Site, Westerstede
- Greece (3):
  - Research Site, Athens
  - Research Site, Ioannina
  - Research Site, Thessaloniki
- Research Site, Guatemala City, Guatemala
- India (10):
  - Research Site, Chenna
  - Research Site, Coimbatore
  - Research Site, Delhi
  - Research Site, Hyderabad
  - Research Site, Kolkata
  - Research Site, Lucknow
  - Research Site, Mangalore
  - Research Site, Mumbai
  - Research Site, New Delhi
  - Research Site, Pune
- Israel (4):
  - Research Site, Ashkelon
  - Research Site, Beer Yaakov
  - Research Site, Jerusalem
  - Research Site, Tel Litwinsky
- Research Site, Roma, Italy
- Mexico (3):
  - Research Site, Guadalajara
  - Research Site, Mexico City
  - Research Site, San Luis Potosí City
- Research Site, Chisinau, Moldova
- Netherlands (2):
  - Research Site, Breda
  - Research Site, Sittard
- New Zealand (3):
  - Research Site, Christchurch
  - Research Site, Grafton
  - Research Site, Hamilton
- Research Site, Skopje, North Macedonia
- Poland (7):
  - Research Site, Bialystok
  - Research Site, Gdansk
  - Research Site, Katowice
  - Research Site, Krakow
  - Research Site, Poznan
  - Research Site, Szczecin
  - Research Site, Warsaw
- Romania (3):
  - Research Site, Bucharest
  - Research Site, Cluj-Napoca
  - Research Site, Timișoara
- Serbia (4):
  - Research Site, Belgrade
  - Research Site, Kragujevac
  - Research Site, Niš
  - Research Site, Novi Sad
- Slovakia (3):
  - Research Site, Bratislava
  - Research Site, Košice
  - Research Site, Martin
- South Africa (3):
  - Research Site, Cape Town
  - Research Site, Durban
  - Research Site, Rosebank
- Switzerland (3):
  - Research Site, Basel
  - Research Site, Sankt Gallen
  - Research Site, Zurich
- Ukraine (6):
  - Research Site, Kharkiv
  - Research Site, Kyiv
  - Research Site, Lviv
  - Research Site, Odesa
  - Research Site, Poltava
  - Research Site, Zaporizhzhya
- United Kingdom (5):
  - Research Site, London
  - Research Site, Newcastle
  - Research Site, Oxford
  - Research Site, Sheffield
  - Research Site, Staffordshire
- Research Site, Vienna, Virgin Islands

REFERENCES:
- [Derived] Gold R, Arnold DL, Bar-Or A, Fox RJ, Kappos L, Chen C, Parks B, Miller C. Safety and efficacy of delayed-release dimethyl fumarate in patients with relapsing-remitting multiple sclerosis: 9 years' follow-up of DEFINE, CONFIRM, and ENDORSE. Ther Adv Neurol Disord. 2020 May 12;13:1756286420915005. doi: 10.1177/1756286420915005. eCollection 2020. PMID 32426039
- [Derived] Mehta D, Miller C, Arnold DL, Bame E, Bar-Or A, Gold R, Hanna J, Kappos L, Liu S, Matta A, Phillips JT, Robertson D, von Hehn CA, Campbell J, Spach K, Yang L, Fox RJ. Effect of dimethyl fumarate on lymphocytes in RRMS: Implications for clinical practice. Neurology. 2019 Apr 9;92(15):e1724-e1738. doi: 10.1212/WNL.0000000000007262. Epub 2019 Mar 27. PMID 30918100
- [Derived] Fox RJ, Gold R, Phillips JT, Okwuokenye M, Zhang A, Marantz JL. Efficacy and Tolerability of Delayed-release Dimethyl Fumarate in Black, Hispanic, and Asian Patients with Relapsing-Remitting Multiple Sclerosis: Post Hoc Integrated Analysis of DEFINE and CONFIRM. Neurol Ther. 2017 Dec;6(2):175-187. doi: 10.1007/s40120-017-0077-5. Epub 2017 Aug 2. PMID 28770420
- [Derived] Fernandez O, Giovannoni G, Fox RJ, Gold R, Phillips JT, Potts J, Okwuokenye M, Marantz JL. Efficacy and Safety of Delayed-release Dimethyl Fumarate for Relapsing-remitting Multiple Sclerosis in Prior Interferon Users: An Integrated Analysis of DEFINE and CONFIRM. Clin Ther. 2017 Aug;39(8):1671-1679. doi: 10.1016/j.clinthera.2017.06.012. Epub 2017 Jul 25. PMID 28751099
- [Derived] Fox RJ, Chan A, Zhang A, Xiao J, Levison D, Lewin JB, Edwards MR, Marantz JL. Comparative effectiveness using a matching-adjusted indirect comparison between delayed-release dimethyl fumarate and fingolimod for the treatment of multiple sclerosis. Curr Med Res Opin. 2017 Feb;33(2):175-183. doi: 10.1080/03007995.2016.1248380. Epub 2016 Nov 10. PMID 27733070
- [Derived] Gold R, Giovannoni G, Phillips JT, Fox RJ, Zhang A, Marantz JL. Sustained Effect of Delayed-Release Dimethyl Fumarate in Newly Diagnosed Patients with Relapsing-Remitting Multiple Sclerosis: 6-Year Interim Results From an Extension of the DEFINE and CONFIRM Studies. Neurol Ther. 2016 Jun;5(1):45-57. doi: 10.1007/s40120-016-0042-8. Epub 2016 Mar 1. PMID 26932146
- [Derived] Giovannoni G, Gold R, Fox RJ, Kappos L, Kita M, Yang M, Sarda SP, Zhang R, Viglietta V, Havrdova E. Relapses Requiring Intravenous Steroid Use and Multiple-Sclerosis-related Hospitalizations: Integrated Analysis of the Delayed-release Dimethyl Fumarate Phase III Studies. Clin Ther. 2015 Nov 1;37(11):2543-51. doi: 10.1016/j.clinthera.2015.09.011. Epub 2015 Oct 31. PMID 26526385
- [Derived] Nakamura K, Brown RA, Narayanan S, Collins DL, Arnold DL; Alzheimer's Disease Neuroimaging Initiative. Diurnal fluctuations in brain volume: Statistical analyses of MRI from large populations. Neuroimage. 2015 Sep;118:126-32. doi: 10.1016/j.neuroimage.2015.05.077. Epub 2015 Jun 3. PMID 26049148
- [Derived] Kita M, Fox RJ, Gold R, Giovannoni G, Phillips JT, Sarda SP, Kong J, Viglietta V, Sheikh SI, Okwuokenye M, Kappos L. Effects of delayed-release dimethyl fumarate (DMF) on health-related quality of life in patients with relapsing-remitting multiple sclerosis: an integrated analysis of the phase 3 DEFINE and CONFIRM studies. Clin Ther. 2014 Dec 1;36(12):1958-1971. doi: 10.1016/j.clinthera.2014.08.013. Epub 2014 Oct 12. PMID 25315404
- [Derived] Fox RJ, Kita M, Cohan SL, Henson LJ, Zambrano J, Scannevin RH, O'Gorman J, Novas M, Dawson KT, Phillips JT. BG-12 (dimethyl fumarate): a review of mechanism of action, efficacy, and safety. Curr Med Res Opin. 2014 Feb;30(2):251-62. doi: 10.1185/03007995.2013.849236. Epub 2013 Oct 22. PMID 24131282
- [Derived] Gold R, Kappos L, Arnold DL, Bar-Or A, Giovannoni G, Selmaj K, Tornatore C, Sweetser MT, Yang M, Sheikh SI, Dawson KT; DEFINE Study Investigators. Placebo-controlled phase 3 study of oral BG-12 for relapsing multiple sclerosis. N Engl J Med. 2012 Sep 20;367(12):1098-107. doi: 10.1056/NEJMoa1114287. PMID 22992073

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were screened and enrolled at 198 investigational sites in 28 countries.
Pre-assignment Details: From screening, 1237 eligible subjects were equally randomized. Of these, 1234 subjects received at least one dose of study treatment and comprised the intent-to-treat (ITT) and safety populations.
Period: Overall Study
Arm/Group | Placebo | BG00012 240 mg Twice Daily (BID) | BG00012 240 mg 3 Times Daily (TID)
Started | 408 (408 participants were dosed; 410 participants were randomized) | 410 (410 participants were dosed; 411 participants were randomized) | 416 (416 participants were dosed; 416 participants were randomized)
Completed | 317 | 315 | 320
Not Completed | 91 | 95 | 96
Not completed — Adverse Event | 22 | 40 | 36
Not completed — Lost to Follow-up | 9 | 11 | 11
Not completed — Withdrawal by Subject | 31 | 22 | 19
Not completed — Physician Decision | 4 | 4 | 3
Not completed — Protocol Violation | 4 | 4 | 8
Not completed — Death | 0 | 0 | 1
Not completed — Other-Unspecified | 21 | 14 | 18

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | BG00012 240 mg Twice Daily (BID) | BG00012 240 mg 3 Times Daily (TID) | Total
Number analyzed (Participants) | 408 | 410 | 416 | 1234
Age, Continuous [Mean (Standard Deviation); unit: Years] | 38.5 (9.14) | 38.1 (9.11) | 38.8 (8.85) | 38.5 (9.03)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 306 | 296 | 306 | 908
  Male | 102 | 114 | 110 | 326
Mean Expanded Disability Status Scale (EDSS) score [Mean (Standard Deviation); unit: units on a scale] — The EDSS scores range from 0.0 (normal exam) to 10.0 (death due to MS).
  units on a scale | 2.48 (1.241) | 2.40 (1.290) | 2.36 (1.188) | 2.42 (1.240)
Mean number of relapses within the previous 3 years [Mean (Standard Deviation); unit: Number of relapses] | 2.5 (1.56) | 2.5 (1.44) | 2.4 (1.27) | 2.5 (1.43)
Mean number of relapses within the past 12 months [Mean (Standard Deviation); unit: Number of relapses] | 1.3 (0.67) | 1.3 (0.67) | 1.3 (0.60) | 1.3 (0.65)
Time since first multiple sclerosis (MS) diagnosis [Mean (Standard Deviation); unit: Years] | 5.8 (5.78) | 5.6 (5.39) | 5.1 (5.29) | 5.5 (5.49)
Mean number of gadolinium (Gd) enhancing lesions [Mean (Standard Deviation); unit: Number of Gd enhancing lesions] — This baseline measure could only be assessed in the magnetic resonance imaging (MRI) cohort. The MRI cohort included 540 intent-to-treat (ITT) subjects who were enrolled at sites that participated in the MRI portion of the study and who had MRI data (180 placebo, 176 BG00012 BID, 184 BG00012 TID). Sites could participate only if their MRI capability was validated by the independent MRI reading center. Approximately 95% of all subjects enrolled at MRI sites participated in the MRI portion of the study.
  Number of Gd enhancing lesions | 1.6 (3.45) | 1.2 (3.30) | 1.2 (4.10) | 1.4 (3.64)

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Subjects Relapsed
Description: A protocol-defined relapse was defined as new or recurrent neurologic symptoms not associated with fever or infection that lasted at least 24 hours, and were separated by at least 30 days from onset of a preceding relapse. All protocol-defined relapses were evaluated by an independent neurolgic evaluation committee. The proportion of subjects with a relapse was estimated using the Kaplan-Meier method, which was based on the time-to-first-relapse survival distribution.
Time Frame: 2 years
Population: The analysis was based on the ITT population, defined as all subjects who were randomized and received at least 1 dose of study medication. Among subjects who switched to an alternative therapy for multiple sclerosis, all the data before the switch were used for the analysis. In all other subjects, all relapses were included in the analysis.
Measure: Number; unit: Proportion of subjects,confirmed relapse
Arm/Group | Placebo | BG00012 240 mg Twice Daily (BID) | BG00012 240 mg 3 Times Daily (TID)
Number analyzed (Participants) | 408 | 410 | 416
Proportion of subjects,confirmed relapse | 0.461 | 0.270 | 0.260

2. Secondary Outcome: Number of New or Newly Enlarging T2 Hyperintense Lesions
Description: The number of new or newly enlarging T2 hyperintense lesions at 2 years that developed in each subject compared to baseline assessed on brain magnetic resonance imaging (MRI) scans. The estimates of mean T2 lesion count were calculated from a negative binomial regression model adjusted for region and baselineT2 lesion volume
Time Frame: 2 years
Population: Of the 540 subjects included in the MRI cohort, 469 subjects (165 placebo, 152 BG00012 BID, 152 BG00012 TID) had post-baseline T2 data and were included in the analysis. Missing data before the use of alternative MS medications and visits after patients switched to alternative MS medications were imputed with the use of a constant rate assumption.
Measure: Mean (95% Confidence Interval); unit: Number of lesions
Groups:
- BG00012 240 mg BID: Participants received two 120 mg BG00012 capsules orally twice daily (BID) and two placebo capsules orally once daily (QD)
- BG00012 240 mg TID: Participants received two 120 mg BG00012 capsules orally three times daily (TID)
Arm/Group | Placebo | BG00012 240 mg BID | BG00012 240 mg TID
Number analyzed (Participants) | 165 | 152 | 152
Number of lesions | 17.0 [12.9 to 22.4] | 2.6 [2.0 to 3.5] | 4.4 [3.2 to 5.9]

3. Secondary Outcome: Number of Gadolinium-enhancing T1-weighted Lesions
Description: The number of Gd-enhancing lesions was assessed using brain MRI scans following administration of gadolinium, a contrast agent. The mean number of Gd-enhancing lesions at 2 years was the average of the number of lesions at 2 years in a treatment group.
Time Frame: 2 years
Population: Of the 540 subjects included in the MRI cohort, 469 (165 placebo,152 BG00012 BID,152 BG00012 TID) had post-baseline Gd-enhancing lesion data & were included in the analysis. Missing data before the use of alternative MS medications & visits after patients switched to alternative MS medications were imputed with the use of a constant rate assumption
Measure: Mean (Standard Deviation); unit: Number of lesions
Arm/Group | Placebo | BG00012 240 mg BID | BG00012 240 mg TID
Number analyzed (Participants) | 165 | 152 | 152
Number of lesions | 1.8 (4.15) | 0.1 (0.63) | 0.5 (1.73)

4. Secondary Outcome: Number of Subjects With Gadolinium (Gd)-Enhancing Lesions
Description: Note: This outcome measure represents the categorical analysis for the previously listed secondary outcome measure "Number of Gadolinium-enhancing T1-weighted lesions"
Time Frame: 2 years
Population: as for outcome 3
Measure: Number; unit: Number of subjects
Arm/Group | Placebo | BG00012 240 mg Twice Daily (BID) | BG00012 240 mg 3 Times Daily (TID)
Number analyzed (Participants) | 165 | 152 | 152
Number of subjects
  0 lesions | 103 | 142 | 130
  1 lesion | 16 | 8 | 10
  2 lesions | 13 | 1 | 2
  3-4 lesions | 15 | 0 | 3
  >=5 lesions | 18 | 1 | 7

5. Secondary Outcome: Annualized Relapse Rate
Description: A protocol-defined relapse was defined as new or recurrent neurologic symptoms not associated with fever or infection that lasted at least 24 hours, and were separated by at least 30 days from onset of a preceding relapse. All protocol-defined relapses were evaluated by an independent neurologic evaluation committee. The adjusted annualized relapse rate was calculated from a negative binomial regression model, adjusted for baseline EDSS (≤ 2.0 vs. >2.0), age (<40 versus ≥40 years), region, and the number of relapses in the 1 year prior to enrollment.
Time Frame: 2 years
Population: The ITT population was defined as all subjects who were randomized and received at least 1 dose of study medication. Among subjects who switched to an alternative therapy for multiple sclerosis, all the data before the switch were used for the analysis. In all other subjects, all relapses were included in the analysis.
Measure: Mean (95% Confidence Interval); unit: Relapses per year
Arm/Group | Placebo | BG00012 240 mg BID | BG00012 240 mg TID
Number analyzed (Participants) | 408 | 410 | 416
Relapses per year | 0.364 [0.303 to 0.436] | 0.172 [0.138 to 0.214] | 0.189 [0.153 to 0.234]

6. Secondary Outcome: Proportion of Subjects Experiencing Progression of Disability Assessed Using the Expanded Disability Status Scale (EDSS)
Description: The EDSS is based on a standardized neurological examination and focuses on symptoms that commonly occur in MS. EDSS scores range from 0.0 (normal) to 10.0 (death due to MS). Disability progression was defined as ≥ 1.0 point increase in subjects with a baseline EDSS of ≥1.0, or a ≥1.5 point increase in subjects with a baseline EDSS = 0, and required that the increase from baseline was confirmed ≥12 weeks later. The proportion of subjects with confirmed (12-week) disability progression was estimated using the Kaplan-Meier method, which was based on the time-to-first-progression survival distribution.
Time Frame: 2 years
Population: The analysis population consisted of the ITT population (all subjects who were randomized and received at least 1 dose of study medication) who had a baseline EDSS assessment. Analysis were based on all observed data. Onset of disability progression must begin before a subject switched to alternative MS medication.
Measure: Number; unit: Proportion of participants
Arm/Group | Placebo | BG00012 240 mg BID | BG00012 240 mg TID
Number analyzed (Participants) | 408 | 409 | 416
Proportion of participants | 0.271 | 0.164 | 0.177

ADVERSE EVENTS:
Time Frame: 2 years
Description: The safety population consisted of all subjects who received at least 1 dose of study treatment. Safety data were analyzed by actual treatment received. Among subjects who switched to an alternative therapy for MS, all the data before the switch were used for the analysis. In all other subjects, all data were included in the analysis.
Groups:
- Total BG00012: Combined BG00012 240 mg twice daily (BID) dose group and BG00012 240 mg 3 times daily (TID) dose group
Arm/Group | Placebo | BG00012 240 mg Twice Daily (BID) | BG00012 240 mg 3 Times Daily (TID) | Total BG00012
Serious Adverse Events (participants affected / at risk) | 86/408 | 74/410 | 65/416 | 139/826
Other Adverse Events (participants affected / at risk) | 384/408 | 394/410 | 393/416 | 787/826
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=408) | BG00012 240 mg Twice Daily (BID) (N=410) | BG00012 240 mg 3 Times Daily (TID) (N=416) | Total BG00012 (N=826)
Gastroenteritis (Infections and infestations) | 0 | 4 | 1 | 5
Pneumonia (Infections and infestations) | 1 | 2 | 0 | 2
Sinusitis (Infections and infestations) | 0 | 1 | 1 | 2
Viral Infection (Infections and infestations) | 0 | 1 | 1 | 2
Appendicitis (Infections and infestations) | 0 | 1 | 0 | 1
H1N1 Influenza (Infections and infestations) | 1 | 0 | 1 | 1
Influenza (Infections and infestations) | 0 | 0 | 1 | 1
Peritonsillar Abscess (Infections and infestations) | 0 | 0 | 0 | 1
Post Viral Fatigue Syndrome (Infections and infestations) | 0 | 1 | 0 | 1
Urinary Tract Infection (Infections and infestations) | 0 | 0 | 1 | 1
Vulval Abscess (Infections and infestations) | 0 | 0 | 1 | 1
Anal Abscess (Infections and infestations) | 1 | 0 | 0 | 0
Diarrhoea Infectious (Infections and infestations) | 1 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0 | 0 | 0
Pelvic Inflammatory Disease (Infections and infestations) | 1 | 0 | 0 | 0
Reiter's Syndrome (Infections and infestations) | 1 | 0 | 0 | 0
Sepsis (Infections and infestations) | 1 | 0 | 0 | 0
Tuberculosis Gastrointestinal (Infections and infestations) | 1 | 0 | 0 | 0
Benign Lung Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 1
Cervix Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1
Neurilemmoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Transitional Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Uterine Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 1 | 1
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Microcytic Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 1 | 1 | 2
Anaphylactoid Reaction (Immune system disorders) | 0 | 0 | 1 | 1
Goitre (Endocrine disorders) | 0 | 1 | 2 | 2
Endocrinopathy Diencephalic (Endocrine disorders) | 0 | 0 | 1 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Adjustment Disorder with Depressed Mood (Psychiatric disorders) | 0 | 1 | 0 | 1
Depression (Psychiatric disorders) | 2 | 1 | 0 | 1
Generalized Anxiety Disorder (Psychiatric disorders) | 0 | 1 | 0 | 1
Mania (Psychiatric disorders) | 0 | 1 | 0 | 1
Narcissistic Personality Disorder (Psychiatric disorders) | 0 | 1 | 0 | 1
Suicidal Ideation (Psychiatric disorders) | 1 | 1 | 0 | 1
Multiple Sclerosis Relapse (Nervous system disorders) | 60 | 39 | 32 | 71
Headache (Nervous system disorders) | 0 | 0 | 2 | 2
Neurological Symptom (Nervous system disorders) | 0 | 1 | 1 | 2
Altered State of Conciousness (Nervous system disorders) | 0 | 0 | 1 | 1
Epilepsy (Nervous system disorders) | 0 | 1 | 0 | 1
Glossopharyngeal Neuralgia (Nervous system disorders) | 0 | 1 | 0 | 1
Ischaemic Stroke (Nervous system disorders) | 0 | 0 | 1 | 1
Multiple Sclerosis (Nervous system disorders) | 0 | 0 | 1 | 1
Transient Global Amnesia (Nervous system disorders) | 0 | 0 | 1 | 1
Transient Ischaemic Attack (Nervous system disorders) | 0 | 1 | 0 | 1
Transverse Sinus Thrombosis (Nervous system disorders) | 0 | 0 | 1 | 1
Viith Nerve Paralysis (Nervous system disorders) | 0 | 1 | 0 | 1
Convulsion (Nervous system disorders) | 1 | 0 | 0 | 0
Encephalopathy (Nervous system disorders) | 1 | 0 | 0 | 0
Grand Mal Convulsion (Nervous system disorders) | 1 | 0 | 0 | 0
Loss of Conciousness (Nervous system disorders) | 1 | 0 | 0 | 0
Migraine (Nervous system disorders) | 1 | 0 | 0 | 0
Restless Legs Syndrome (Nervous system disorders) | 1 | 0 | 0 | 0
Vertigo Positional (Ear and labyrinth disorders) | 0 | 0 | 1 | 1
Acute Coronary Syndrome (Cardiac disorders) | 0 | 0 | 1 | 1
Cardiac Failure (Cardiac disorders) | 0 | 0 | 1 | 1
Cardiac Failure Congestive (Cardiac disorders) | 0 | 0 | 1 | 1
Flushing (Vascular disorders) | 0 | 1 | 1 | 2
Varicose Vein (Vascular disorders) | 0 | 1 | 1 | 2
Deep Vein Thrombosis (Vascular disorders) | 0 | 0 | 1 | 1
Peripheral Ischaemia (Vascular disorders) | 1 | 0 | 0 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 0 | 3 | 3
Vomiting (Gastrointestinal disorders) | 0 | 1 | 1 | 2
Abdominal Hernia (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Abdominal Pain Lower (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Gastrontestinal Disorder (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Hiatus Hernia (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Colitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Colitis Ulcerative (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Peritoneal Haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0 | 1
Hepatitis Cholestatic (Hepatobiliary disorders) | 0 | 1 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
Stevens-Johnson Syndrome (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Dermatitis Allergic (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Sjogren's Syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Polyarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Synovial Cyst (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Renal Colic (Renal and urinary disorders) | 0 | 0 | 1 | 1
Ureterocele (Renal and urinary disorders) | 0 | 1 | 0 | 1
Ovarian Cyst (Reproductive system and breast disorders) | 1 | 1 | 2 | 3
Adenomyosis (Reproductive system and breast disorders) | 0 | 0 | 1 | 1
Endometriosis (Reproductive system and breast disorders) | 0 | 1 | 0 | 1
Ovarian Cyst Ruptured (Reproductive system and breast disorders) | 0 | 1 | 0 | 1
Menstrual Disorder (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Pelvic Pain (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Uterine Haemorrhage (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Hydrocele (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 1
Pyrexia (General disorders) | 0 | 1 | 1 | 2
Non-Cardiac Chest Pain (General disorders) | 0 | 0 | 1 | 1
Influenza Like Illness (General disorders) | 1 | 0 | 0 | 0
Pelvic Mass (General disorders) | 1 | 0 | 0 | 0
Allergy Test (Investigations) | 0 | 0 | 1 | 1
Blood Glucose Increased (Investigations) | 0 | 0 | 1 | 1
Colonoscopy (Investigations) | 0 | 1 | 0 | 1
Investigation (Investigations) | 0 | 0 | 1 | 1
Medical Observation (Investigations) | 0 | 0 | 1 | 1
Hepatic Enzyme Increased (Investigations) | 1 | 0 | 0 | 0
Road Traffic Accident (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 2
Ankle Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Concussion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Meniscus Lesion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Postoperative Fever (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Procedural Hypotension (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Radius Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Traumatic Brain Injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Wrist Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Femoral Neck Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Tendon Rupture (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0
Tibia Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Female Sterilization (Surgical and medical procedures) | 0 | 1 | 0 | 1
Hysterectomy (Surgical and medical procedures) | 0 | 1 | 0 | 1
Venous Stent Insertion (Surgical and medical procedures) | 0 | 0 | 1 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=408) | BG00012 240 mg Twice Daily (BID) (N=410) | BG00012 240 mg 3 Times Daily (TID) (N=416) | Total BG00012 (N=826)
NASOPHARYNGITIS (Infections and infestations) | 101 | 108 | 109 | 217
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 53 | 63 | 51 | 114
URINARY TRACT INFECTION (Infections and infestations) | 53 | 55 | 54 | 109
INFLUENZA (Infections and infestations) | 39 | 34 | 48 | 82
SINUSITIS (Infections and infestations) | 20 | 17 | 34 | 51
BRONCHITIS (Infections and infestations) | 18 | 21 | 26 | 47
GASTROENTERITIS (Infections and infestations) | 21 | 26 | 20 | 46
RHINITIS (Infections and infestations) | 19 | 12 | 16 | 28
DEPRESSION (Psychiatric disorders) | 32 | 29 | 33 | 62
INSOMNIA (Psychiatric disorders) | 19 | 20 | 20 | 40
MULTIPLE SCLEROSIS RELAPSE (Nervous system disorders) | 181 | 109 | 107 | 216
HEADACHE (Nervous system disorders) | 80 | 81 | 78 | 159
PARAESTHESIA (Nervous system disorders) | 38 | 35 | 38 | 73
HYPOAESTHESIA (Nervous system disorders) | 27 | 20 | 24 | 44
DIZZINESS (Nervous system disorders) | 23 | 19 | 22 | 41
VERTIGO (Ear and labyrinth disorders) | 15 | 13 | 29 | 42
FLUSHING (Vascular disorders) | 20 | 153 | 132 | 285
HOT FLUSH (Vascular disorders) | 8 | 31 | 29 | 60
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 19 | 25 | 21 | 46
COUGH (Respiratory, thoracic and mediastinal disorders) | 18 | 22 | 19 | 41
DIARRHEA (Gastrointestinal disorders) | 55 | 62 | 78 | 140
NAUSEA (Gastrointestinal disorders) | 38 | 53 | 54 | 107
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 28 | 40 | 52 | 92
ABDOMINAL PAIN (Gastrointestinal disorders) | 22 | 46 | 37 | 83
VOMITING (Gastrointestinal disorders) | 24 | 40 | 29 | 69
DYSPEPSIA (Gastrointestinal disorders) | 12 | 23 | 24 | 47
CONSTIPATION (Gastrointestinal disorders) | 19 | 14 | 18 | 32
GASTROINTESTINAL DISORDER (Gastrointestinal disorders) | 6 | 9 | 20 | 29
PRURITIS (Skin and subcutaneous tissue disorders) | 19 | 42 | 33 | 75
RASH (Skin and subcutaneous tissue disorders) | 13 | 34 | 27 | 61
ERYTHEMA (Skin and subcutaneous tissue disorders) | 5 | 20 | 33 | 53
BACK PAIN (Musculoskeletal and connective tissue disorders) | 57 | 59 | 46 | 105
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 39 | 46 | 37 | 83
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 29 | 37 | 29 | 66
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 20 | 13 | 27 | 40
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 26 | 12 | 14 | 26
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 21 | 11 | 10 | 21
PROTEINURIA (Renal and urinary disorders) | 34 | 38 | 50 | 88
HAEMATURIA (Renal and urinary disorders) | 19 | 26 | 26 | 52
MICROALBUMINURIA (Renal and urinary disorders) | 11 | 21 | 17 | 38
FATIGUE (General disorders) | 54 | 57 | 63 | 120
PYREXIA (General disorders) | 21 | 16 | 18 | 34
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 13 | 29 | 27 | 56
ALBUMIN URINE PRESENT (Investigations) | 12 | 24 | 22 | 46

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The provisions of the agreements are subject to confidentiality but generally the PI can publish, for noncommercial purposes only, results and methods of the trial, but no other Sponsor Confidential Information. PI must give Sponsor no less than 60 days to review any manuscript for a proposed publication and must delay publication for up to 90 days thereafter if Sponsor needs to file any patent application to protect any of Sponsor's intellectual property contained in the proposed publication.